CLINICAL TRIAL: NCT02378662
Title: Safety & Efficacy of Prolonged Physiologic Erythropoietin (EPO) Level Treatment of Anemia in End Stage Renal Disease (ESRD) Patients Undergoing Peritoneal Dialysis (PD)Using MDGN201 TARGTEPO
Brief Title: TARGTEPO Treatment for Anemia in End Stage Renal Disease (ESRD) Patients Undergoing Peritoneal Dialysis (PD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's decision of the Early Termination of the study.
Sponsor: Aevi Genomic Medicine, LLC, a Cerecor company (Industry)
Collaborators: Medgenics Medical Israel Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MG-EP-RF-03
Record Dates: First submitted 2015-02-22; First posted 2015-03-04 (Estimated); Results first posted 2018-10-19 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2017-12

CONDITIONS: Anemia of End Stage Renal Disease
Keywords: Peritoneal Dialysis; End Stage Renal Disease; Anemia
MeSH Terms: conditions — Kidney Failure, Chronic; Anemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): MDGN201 TARGTEPO secreting EPO (18-25 IU/Kg/day)
  Interventions: Biological: MDGN201 TARGTEPO
- Group B (Experimental): MDGN201 TARGTEPO secreting EPO (35-45 IU/Kg/day)
  Interventions: Biological: MDGN201 TARGTEPO

INTERVENTIONS:
Biological: MDGN201 TARGTEPO — MDGN201 TARGTEPO secreting EPO

SUMMARY:
The objectives of this study are to assess safety and to evaluate the biologic activity of TARGTEPO treatment in Peritoneal Dialysis patients

DETAILED DESCRIPTION:
This is a Phase II, open-label study. Each patient will receive targeted dose of Erythropoietin (EPO) delivered via TARGTEPO.

The targeted doses will be determined according to 2 cohorts as follows: Group A (18-25 IU/Kg/day), Group B (35-45 IU/Kg/day). The objective is to evaluate safety and biologic activity of TARGTEPO treatment when maintaining Hb levels within the target range of 9-12 g/dl. Biological activity assessments will include duration of TARGTEPO secretion as measured by serum EPO levels above baseline.

ELIGIBILITY:
Inclusion Criteria:

1. Subject diagnosed with Anemia due to Chronic Renal Failure CKD stage 5 on peritoneal dialysis treatment for at least 6 months. Average Hb during last month between 9 to 12g/dL.
2. Kt/V >1.
3. INR ≤1.2
4. Serum albumin >3.2
5. Subjects with adequate iron stores (transferrin saturation > 20.0% and/or ferritin >100 ng/ml).

Exclusion Criteria:

1. Uncontrolled hypertension (defined as diastolic blood pressure > 110 mmHg or systolic blood pressure > 180 mmHg during screening).
2. Subjects who receive oral anti-coagulation treatment (e.g. warfarin)
3. Subjects who receive Acetyl Salicylic Acid (ASA) above 325 mg/day or patients who receive ASA treatment between 100mg/d and 325 mg/d who cannot discontinue it for 1 week prior to each Harvest or Implantation procedure
4. Congestive heart failure (New York Heart Association functional class III or IV).
5. Grand mal seizures within 2 years of the screening visit.
6. Clinical evidence of severe hyperparathyroidism as defined by PTH levels of > 10 times the upper normal limits.
7. Major surgery within 12 weeks of the screening visit.
8. Systemic hematologic diseases (e.g., sickle cell anemia, thalassemia (excluding Thalassemia minor), myelodysplastic syndromes, hematologic malignancy, myeloma, hemolytic anemia).
9. Current systemic infection, active inflammatory disease, or malignancy under active treatment.
10. Subjects known to have tested positive at any time in the past for antibodies to erythropoietic proteins.
11. Subject has history of malignancy within the past 2 years prior to the screening visit, with the exception of basal cell carcinoma.
12. Subjects with other concurrent severe and/or uncontrolled medical condition which could compromise participation in the study (i.e. active infection, uncontrolled diabetes, uncontrolled hypertension, congestive heart failure, unstable angina, ventricular arrhythmias, active ischemic heart disease, myocardial infarction within six months, uncompensated cirrhosis, active upper GI tract ulceration).
13. Subject is currently enrolled in, or has not yet completed a period of at least 30 days or five half-lives of the investigational drug whichever is longer, since ending other investigational device or drug trial(s) prior to Screening phase.
14. Psychiatric, addictive, or any other disorder that compromises ability to provide informed consent for participation in this study.
15. Female subjects of child-bearing potential and males that do not agree to use acceptable methods of contraception during the study.
16. Pregnant and lactating female subjects.
17. Chronic alcoholic or drug abuse subjects.
18. Steroid or other immunosuppressive treatment (other than topical or inhaled steroids).
19. Subjects unwilling or unable to comply with the study procedures.
20. EPO Naïve subjects.
21. Known sensitivity to Gentamycin and Amphotericin
22. History of chronic or active Hepatitis B and/or C infection or positive serology at screening and known positive HIV or positive serology at screening.
23. Subject had blood transfusion within 84 days prior to Screening visit.
24. Subject has a date for renal transplantation.
25. Refer to the USPI - Depo-Medrol - Methylprednisolone Acetate - Injectable (Appendix A) for any concomitant drug taken by the patient which its interaction with Depo-Medrol will warrant exclusion from this protocol.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-04; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shany Blum, MD PhD, Study Director — Medgenics Medical Israel Ltd.
Locations (2):
- Israel (2):
  - Barzili Medical Center, Ashkelon
  - Assaf Harofeh Medical Center, Zrifin

IPD SHARING:
Plan to Share IPD: No
Early phase and small feasibility study.

RESULTS

PARTICIPANT FLOW:
Groups:
- Group A: 18-25 IU/Kg/day
- Group B: 35-45 IU/Kg/day
Period: Overall Study
Arm/Group | Group A | Group B
Started | 2 | 0
Harvesting | 2 | 0
Implantation | 2 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Early Discontinuation | 2 | 0

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 0 | 2
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Patients Who Achieved Biological Activity of MDGN201 TARGTEPO Secretion as Measured by Serum Erythropoietin (EPO) Levels Above Baseline
Time Frame: 52 weeks
Population: No statistical analysis was performed as only two subjects were treated with MDGN201 TARGTEPO due to Sponsor's decision to discontinue study.
Measure: Count of Participants; unit: Participants
Arm/Group | Group A | Group B
Number analyzed (Participants) | 2 | 0
Participants | 2 | 0

ADVERSE EVENTS:
Arm/Group | Group A | Group B
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 2/2 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group A (N=2) | Group B (N=0)
Intermittent Muscle cramps in both legs (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Catheter exit site infection (Infections and infestations) | 1 (1) | 0 (0)
Allergic reaction to ciprofloxacin (Immune system disorders) | 1 (1) | 0 (0)
Swelling in right groin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Redness in right groin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Should the investigator wish to publish the results of this study, the investigator agrees to provide Medgenics with a manuscript for review 60 days prior to submission for publication. Medgenics retains the right to delete from the manuscript information that is confidential and proprietary and to object to suggested publication and/or its timing (at the Company's sole discretion).